CLINICAL TRIAL: NCT04839081
Title: Neuropathic Characteristics of Rheumatoid Hand Pain and it's Relation to Sensory Thresholds and Sleep Quality: a Case-control Study
Brief Title: Neuropathic Hand Pain in Rheumatoid Arthritis
Status: Active, not recruiting | Type: Observational
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Taciser Kaya, Associate professor, MD, Bozyaka Training and Research Hospital
Other Study IDs: 45986TK
Record Dates: First submitted 2021-04-08; First posted 2021-04-09 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Surveys and Questionnaires; Equipment and Supplies; Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- RA patients: RA patients diagnosed according to the 1987 ACR Criteria
  Interventions: Other: questionnaires and inventories
- Control: Age- and sex-matched control subjects with nociceptive/mechanical pain complaint other than in hand, lasting more than three months
  Interventions: Other: questionnaires and inventories

INTERVENTIONS:
Other: questionnaires and inventories — questionnaires and inventories related to primary end secondary outcomes will be applied and physical examination will be performed.
  Other Names: physical examination

SUMMARY:
Investigators have aimed to estimate prevalence of neuropathic hand pain in RA patients and it's relation with sleep quality and sensory thresholds. For this purpose a case-control study design was planned. Age- and sex-matched control subjects will be chosen among individuals submitted to out-patient clinic with the complaint of nociceptive/mechanical pain other than in hand, lasting more than three months

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic, inflammatory rheumatic disease that predominantly affecting peripheral joints. Patients with RA are suffered from severe hand pain and functional loss because of synovitis in hand joints. The fact that patients with low disease activity may complain from hand pain suggests that pain is mediated by mechanisms other than inflammation. Contribution of central sensitization to pain sensation of RA patients is of interest currently. Several authors reported the neuropathic characteristics of hand pain in RA. Hand pain is primarily nociceptive in RA patients but the possibility of variances in cutaneous sensitivity due to nociceptive input from joints has been suggested. Increased sensitivity with light touch has been demonstrated over hands of RA patients. In RA patients, alterations in central processing of somatosensory function and allodynia over inflamed joints have been reported. Poor sleep quality is another issue for RA patients and it's association with pain was reported. However impact of neuropathic hand pain on sleep quality was not understood exactly probably due to the scarce of the studies investigating this association. Also, to the best of investigators' knowledge, the relation between neuropathic component of pain and sensory threshold alterations in rheumatoid hand was not studied to date.

So, investigators have aimed to estimate prevalence of neuropathic hand pain in RA patients and it's relation with sleep quality and sensory thresholds. For this purpose a case-control study design was planned. Age- and sex-matched control subjects will be chosen among individuals submitted to out-patient clinic with nociceptive/mechanical pain complaint other than in hand lasting more than three months. Also whether sensory thresholds in rheumatoid hands differ from healthy hands will be assessed. Participants in control group will be subjected to same exclusion criteria too.

This design will allow the investigators to determine whether hand pain in RA patients displays neuropathic character more frequently than any other chronic nociceptive pain does. Moreover, it will be possible to compare sensory thresholds between healthy and rheumatoid hand. RA patients diagnosed according to the 1987 American College of Rheumatology criteria will be recruited. Demographics and disease related variables will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Being diagnosed with RA according to the 1987 ACR Criteria
2. Visual Analogue Scale hand pain score ≥ 3

Exclusion Criteria:

1. Diabetes mellitus, renal insufficiency, hypothyroidism
2. Carpal tunnel syndrome, postherpetic neuralgia, cervical spinal cord compression
3. Cervical radiculopathy
4. Fibromyalgia
5. Malignancy
6. Hand muscle weakness of even one grade on Medical Research Council Manual Muscle Testing scale
7. Upper motor neuron sign on physical examination of hands
8. Pregnancy
9. In the last three months medical treatment leading to neuropathy (colchicine etc.)
10. In the last three months drug use for the treatment of fibromyalgia, depression or anxiety

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA patients having hand pain with severity of 3 or more on 100 mm VAS and age- and sex-matched control subjects will be chosen among individuals submitting to our out-patient clinic with nociceptive/mechanical pain complaint lasting more than three months
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Neuropathic pain | Once, at baseline
  It will be assessed using the painDETECT questionnaire. This questionnaire, contains nine questions all of which are selfreport. Seven items are rated on a six point Likert scale and thus are scored between 0-5. These seven questions query some sensations such as burning, tingling or prickling, allodynia, numbness etc. Apart from these seven items, one item assesses the radiation of pain and the other one item looks for the temporal characteristics of pain. A total score of 12 or less indicates neuropathic component is unlikely, 13-18 means possible neuropathic component and19 or greater means a neuropathic component is likely. Beside these, there are three items in a separate section measuring severity of pain at the time of evaluation, on average and maximum over the past month. This section is not taken into account in scoring
Sleep quality | Once, at baseline
  It will be assessed using Pittsburgh Sleep Quality Index (PSQI). It was developed by Buysse and coworkers in 1989.
  This index measures sleep quality quantitatively and covers 24 questions. Nineteen questions are self-rated and scoring is based on these self-rated questions, other five questions that rating by partner are not taken into account while calculating total score. Questionnaire measures seven domains; subjective sleep quality (question 6), sleep latency (question 2 and 5a), sleep duration (question 4), habitual sleep efficiency (question 1,3,4), sleep disturbances (question 5b-j), use of sleep medication (question 7), and daytime dysfunction (question 8 and 9) over the last month.
  Seven domain scores give a result on a 0 to 3 scale. To yield a total score the domain scores are summed. Total score varies between 0 and 21. Higher scores indicate worse sleep quality.

SECONDARY OUTCOMES:
Light touch-pressure threshold | Once, at baseline
  It will be assessed using Semmes-Weinstein monofilament test composing of five filaments ranging in thickness from 2.83 to 6.65 mm and applying force ranging from 0.07 g to 300 g. The procedure is started by getting the thinnest filament in contact to relevant skin region. If it is not felt after three trials with same filament, examiner proceeds with the next more larger filament until touch felt by the patient.
Depression | Once, at baseline
  It will be assessed using Beck Depression Inventory. It is is a 21-question multiple-choice self-report inventory quantifies the symptoms of depression. Each question is rated between 0 and 3 to reflect the intensity of statements. All points are summed arithmetically to obtain a total score which ranges between 0 and 63. Higher scores indicate more intense depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Taciser Kaya, Assoc. prof, Principal Investigator — Izmir Bozyaka Training and Reseach Hospital
Locations (1):
- Izmir Bozyaka Training and Research Hospital, Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] Koop SM, ten Klooster PM, Vonkeman HE, Steunebrink LM, van de Laar MA. Neuropathic-like pain features and cross-sectional associations in rheumatoid arthritis. Arthritis Res Ther. 2015 Sep 3;17(1):237. doi: 10.1186/s13075-015-0761-8. PMID 26335941
- [Background] Joharatnam N, McWilliams DF, Wilson D, Wheeler M, Pande I, Walsh DA. A cross-sectional study of pain sensitivity, disease-activity assessment, mental health, and fibromyalgia status in rheumatoid arthritis. Arthritis Res Ther. 2015 Jan 20;17(1):11. doi: 10.1186/s13075-015-0525-5. PMID 25600850
- [Background] Loppenthin K, Esbensen BA, Jennum P, Ostergaard M, Tolver A, Thomsen T, Midtgaard J. Sleep quality and correlates of poor sleep in patients with rheumatoid arthritis. Clin Rheumatol. 2015 Dec;34(12):2029-39. doi: 10.1007/s10067-015-2875-4. Epub 2015 Jan 27. PMID 25620673
- [Background] Ulus Y, Akyol Y, Tander B, Durmus D, Bilgici A, Kuru O. Sleep quality in fibromyalgia and rheumatoid arthritis: associations with pain, fatigue, depression, and disease activity. Clin Exp Rheumatol. 2011 Nov-Dec;29(6 Suppl 69):S92-6. Epub 2012 Jan 3. PMID 22243555